CLINICAL TRIAL: NCT06231342
Title: Endotracheal Tube (ETT) 180: Stylet-loaded Endotracheal Tube Rotation Before Insertion to Decrease the Risk of Postoperative Sore Throat: a Randomized Double-Blind Prospective Trial.
Brief Title: Endotracheal Tube (ETT) 180: Stylet-loaded Endotracheal Tube Rotation Before Insertion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Suren Soghomonyan, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022H0220
Record Dates: First submitted 2024-01-12; First posted 2024-01-30 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia, Endotracheal

STUDY DESIGN:
Intervention Model Description: A prospective double-blinded randomized trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects and research personnel assessing subjects during follow-ups will be blinded throughout the study. Only the clinicians inside the operative room will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Direct Laryngoscopy (DL) (Active Comparator): Standard laryngoscope use to insert the endotracheal tube and removing the stylet without any rotation.
  Interventions: Device: Direct Laryngoscope (DL)
- Direct laryngoscopy (DLE) plus Endotracheal Tube (ETT) 180 maneuver (Active Comparator): Standard laryngoscope use to insert the endotracheal tube and removing the stylet using a 180-degree rotation.
  Interventions: Device: Direct Laryngoscope (DL); Procedure: Endotracheal Tube (ETT) 180
- Video laryngoscopy plus Endotracheal Tube (ETT) 180 maneuver (VLE) (Active Comparator): Video laryngoscope use to insert the endotracheal tube and removing the stylet using a 180-degree rotation.
  Interventions: Device: Video laryngoscope (VL); Procedure: Endotracheal Tube (ETT) 180

INTERVENTIONS:
Device: Direct Laryngoscope (DL) — DL allows visualization of the larynx. It is used during general anesthesia, for surgical procedures of the larynx, and during resuscitation.
  Arms: Direct Laryngoscopy (DL); Direct laryngoscopy (DLE) plus Endotracheal Tube (ETT) 180 maneuver
Device: Video laryngoscope (VL) — VL facilitates intubation while allowing clinicians to share and record real-time high-resolution images and video.
  Arms: Video laryngoscopy plus Endotracheal Tube (ETT) 180 maneuver (VLE)
Procedure: Endotracheal Tube (ETT) 180 — A novel maneuver has been described to decrease the insult from stylet named Endotracheal Tube (ETT) 180; a clockwise rotation of the stylet-loaded Endotracheal Tube (ETT) 180 degrees on its axis right after the tip of Endotracheal Tube (ETT) passes the patient's vocal cords (glottis) before fully inserting the Endotracheal Tube (ETT) and then, pulling the stylet out. This maneuverer allows the stylet to match the posterior angulation of the trachea.
  Arms: Direct laryngoscopy (DLE) plus Endotracheal Tube (ETT) 180 maneuver; Video laryngoscopy plus Endotracheal Tube (ETT) 180 maneuver (VLE)

SUMMARY:
The main objective of the proposed study is to clarify whether rotating a stylet-loaded endotracheal tube (ETT) 180 degrees prior to intubation will decrease the incidence of postoperative throat soreness, when compared to standard technique used in Standard of Care.

DETAILED DESCRIPTION:
The researcher who is not blinded will randomize the patient to one of the three groups.

Specific technique and procedure:

* Investigators anesthesiologists assigned to perform the laryngoscopies will be limited to 6 with minimum 2 years of attending experiences to balance the variability. The results of inter-operator bias will be analyzed.
* Endotracheal Tube (ETT) size will be: 7.0 for men and women unless there will be clinical indications to use a different size of Endotracheal Tube.
* Stylet preparation: 75-degree angulation shaped preoperatively and ready for use
* Blade for either McGrath, Macintosh, or direct laryngoscopy will be size 3 for women and size 4 for men.
* Endotracheal Tube (ETT) 180: inserting endotracheal tube loaded with stylet, rotating the tube 180 degree clockwise as soon as the tube tip passes the vocal cords (glottis), and removing the stylet after the tube cuff passes through the vocal cords, which is a common practice.
* Endotracheal Tube cuff filling air pressure will be 20 cmH2O. Inflation will be made using a hand-held airway pressure manometer.
* Patient's data collection will be blinded for both patient and Investigators anesthesiologists assigned to perform the laryngoscopies
* No medications including opiates, monitoring options, and medical decisions will be altered by the study.

A member of the research team will follow-up (in person or phone-call) with each patient in the Post Anesthesia Care Unit (PACU) and 24+/- 3 hours after endotracheal tube removal to collect information regarding any symptoms of hoarseness or sore throat.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - III
* Ambulatory patients undergoing general anesthesia with an Endotracheal Tube (ETT) placement
* Admitted patients undergoing general anesthesia an Endotracheal Tube (ETT) placement
* Age > 18 and < 90 years old
* BMI < 50

Exclusion criteria:

* Age < 18 years old or age > 90 years old
* Pregnant women
* Prisoners
* Any surgery involving the pharynx, larynx, vocal cords, trachea that will create confounding factors related to postoperative sore throat
* History of difficult airway
* Critically ill patients requiring intensive care

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative sore throat | 24 hours after Endotracheal Tube (ETT) placement
  To assess the differences in incidence of postoperative sore throat after intubation between the conventional technique and ETT 180 rotation of the ETT.

SECONDARY OUTCOMES:
Incidence of hoarseness/sore throat | 24 hours after Endotracheal Tube (ETT) placement
  To assess the incidence of hoarseness/sore throat
Severity of hoarseness/sore throat | 24 hours after Endotracheal Tube (ETT) placement
  To assess the severity of hoarseness/sore throat using a 0-3-point scale (units), where 0 = no hoarneseness/sore throat at all and and 3 = very bad hoarseness/sore throat sensation.
Incidence of analgesic medication requirements to treat sore throat. | 24 hours after Endotracheal Tube (ETT) placement
  To assess the incidence of analgesic medication to treat sore throat sensation.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided